CLINICAL TRIAL: NCT00797160
Title: Propofol and Remifentanil Versus Midazolam and Remifentanil as Premedication Allowing Very Early Extubation After Surfactant Treatment in Preterm Neonates With Respiratory Distress Syndrome
Brief Title: Propofol Versus Midazolam as Premedication for Preterm Neonates With Respiratory Distress Syndrome (RDS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Yerkes Pereira e Silva, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0011.0.287.000-08
Record Dates: First submitted 2008-11-20; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: propofol; midazolam; neonate; tracheal intubation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: propofol — 2mg/Kg IV in bolus before tracheal intubation

SUMMARY:
The aim of the study is to compare the intubation conditions among propofol and remifentanil versus midazolam and remifentanil in premature neonates with respiratory distress syndrome. At the same time, to show the group of drugs that could let the neonates with no residual sedation after the use of surfactant (the possibility of the premature neonates to be readily extubated after the use of surfactant).

DETAILED DESCRIPTION:
It has been demonstrated that remifentanil, due to it its very short context-sensitive, has an interesting potential for use in premature neonates with respiratory distress syndrome. Indeed, remifentanil allowed an adequate level of sedation and analgesia as well as rapid recovery after discontinuation. The aim of the present study was to compares the intubation conditions among propofol and remifentanil versus midazolam and remifentanil in premature neonates with respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28-34 wk
* Clinical and radiological features compatible with respiratory distress syndrome that required elective tracheal intubation and surfactant therapy
* Hemodynamic stability before tracheal intubation
* Signature (parents) consent form

Exclusion Criteria:

* The presence of major congenital malformations
* Birth weigh less than 1000 g
* Previous use of opioid or other sedative drug for any reason
* Previous tracheal intubation
* Hemodynamic instability before the indication of tracheal intubation
* Refuse of the parents to enroll the neonate in the study protocol

Ages: 30 Minutes to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Time until extubation after bolus dose as premedication for tracheal intubation | within the first 3 days of life

SECONDARY OUTCOMES:
Quality of intubation with the combination of drugs used for premedication | within the first 2 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Yerkes P Silva, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Department of Neonatology of Julia Kubitschek Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] SILVA,Y.P. et al. Morphine versus remifentanil for intubating preterm neonates. Short report.Archives of Disease in Childhood Fetal & Neonatal Edition;92:4.2007. Dani C, Bertini G, Pezzati M, et al. Early Extubation and Nasal Continuous Positive Airway Pressure After Surfactant Treatment for Respiratory Distress Syndrome Among Preterm Infants <30 Weeks' Gestation. Pediatrics 2004; 113:560-563. Carbajal R, Eble B, Anand KJS. Premedication for Tracheal Intubation in Neonates: Confusion or Controversy? Seminars in Perinatology 2007; 31:309-317. Silva YP, Gomez RS, Marcatto JO, et al. Early awakening and extubation with remifentanil in ventilated premature neonates. Pediatric Anesthesia 2008; 18:176-183. Welzing L, Roth B. Experience with remifentanil in neonates and infants. Drugs 2006; 66(10):1339-1350.